CLINICAL TRIAL: NCT00439868
Title: A Cross-over Study to Evaluate the Effect of WELLBUTRIN XL on Intraocular Pressure in Healthy Volunteers
Brief Title: A Study To Evaluate The Effect Of WELLBUTRIN XL On Intraocular Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Purpose: Diagnostic
Other Study IDs: WXL108709
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Depressive Disorder
Keywords: WELLBUTRIN XL, intraocular pressure, healthy volunteers
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group 1 (Experimental): Subjects in Period 1 of treatment group 1 will receive oral doses of extended release WELLBUTRIN XL tablets for 2 weeks, from Days 1-3 subject will receive 150 milligram (mg) tablets once daily (QD) and from Days 4-14 300 mg QD. In Period 2 subject will receive placebo for 2 weeks.
  Interventions: Drug: WellbutrinXL; Drug: placebo
- Treatment Group 2 (Experimental): Subjects in Period 1 of Treatment group 2 will receive Placebo for 2 weeks and in Period 2 subject will receive oral doses of extended release WELLBUTRIN XL for 2 weeks, from Days 1-3 subject will receive 150 milligram (mg) tablets once daily (QD) and from Days 4-14 300 mg QD.
  Interventions: Drug: WellbutrinXL; Drug: placebo

INTERVENTIONS:
Drug: WellbutrinXL — WELLBUTRIN XL tablets will be available with dose strength of 150 and 300 mg.
Drug: placebo — Matching placebo tablets to WELLBUTRIN XL.
  Other Names: WellbutrinXL

SUMMARY:
This study will be conducted in healthy volunteers to investigate the effect on intraocular pressure of 2 weeks of treatment with 300mg WELLBUTRIN XL/day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females.
* Non-smokers
* Agree to remain in the clinic for the time defined in the protocol.
* Normal ECG.

Exclusion Criteria:

* Any serious medical disorder or condition.
* Any history of an endocrine disorder.
* Any clinically significant laboratory abnormality.
* History of psychiatric illness.
* Any history of suicidal attempts or behavior.
* Risk factors for precipitation of angle closure glaucoma or elevated IOP.
* Inability to refrain from use of contact lenses during the study days, if correction is required.
* Self-administered Beck Depression Inventory II scale total score greater than 9, and a suicide question score of greater than zero.
* Current or past history of seizure disorder or brain injury (traumatic or disease-related); or any condition which, in the opinion of the investigator, predisposes to seizure - Women having a positive serum HCG pregnancy test at screening, a positive urine pregnancy test before admission to the Unit during the in-house periods, who are not willing to use acceptable methods of contraception or who are lactating or planning to become pregnant within the three months following the screening visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2007-02-16 (Actual); Primary Completion 2007-06-08 (Actual); Study Completion 2007-06-08 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure at Day -1, Days 1 & 14. | at Day -1, Days 1 & 14.

SECONDARY OUTCOMES:
Intraocular pressure,Pupil diameter, anterior chamber angle | Days-1,1&14
Wellbutrin XL plasma level | Days1,12-14
adverse events | each visit
lab tests,ECG,vital signs: | screening,followup
lab tests: | Days-2,13-14
ECG: | Day 14
vital signs: | Days-2,-1,1,14

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Gainesville, Florida, United States

REFERENCES:
- See also: Results for study WXL108709 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/WXL108709?search=study&search_terms=WXL108709#rs